CLINICAL TRIAL: NCT01366469
Title: Inflammatory Biomarkers Predict Pulmonary Outcomes in Coronary Artery Bypass Grafting
Acronym: CABG BALF
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Omar Lattouf, Professor of Surgery, Emory University
Other Study IDs: IRB00046469; CABG BALF (Other: Other)
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Coronary Artery Disease; Chronic Obstructive Pulmonary Disease
Keywords: coronary artery bypass grafting; coronary artery disease; chronic obstructive pulmonary disease
MeSH Terms: conditions — Coronary Artery Disease; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — BAL fluid, Serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary objective of this pilot study is to identify and quantify inflammatory and genetic markers from bronchoalveolar lavage fluid (BALF) and serum in patients with a history of chronic obstructive pulmonary disease (COPD) undergoing elective coronary revascularization (CABG) to determine the risk of developing post operative respiratory failure. To achieve this objective, this proposal outlines the following specific aims:

Aim #1. To identify from BALF and serum, the change in inflammatory and genetic markers in patients with a history of COPD undergoing CABG. BALF and serum samples will be obtained at the time of intubation immediately prior to surgery and again upon skin closure immediately after the surgical procedure.

Aim #2. To determine the extent to which inflammatory and/or genetic markers correlate with post-operative pulmonary complications defined as prolonged mechanical ventilation (> 24 hours), pneumonia, and/or tracheostomy.

Aim #3. To inform the development and implementation of a large pivotal trial which may impact clinical decision-making during the initial pre-operative outpatient assessment of COPD patients undergoing CABG.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective CABG
* Current diagnosis of COPD
* Ability to provide signed informed consent to participate
* > 18 years of age

Exclusion Criteria:

* Concomitant valve surgery
* Urgent or emergent coronary surgery
* Current steroid therapy
* Active smoker and/or positive urine co-nicotine

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from Cardiothoracic surgery service
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure | During Hospitalization
  The identification of specific inflammatory and genetic markers associated with post-operative pulmonary complications in this population of elective CABG patients with a history of COPD.

SECONDARY OUTCOMES:
Secondary outcome measure | 30 Day Follow-up
  Post-operative pulmonary complications: prolonged mechanical ventilation (defined as >24 hours), atelectasis, pneumonia, exacerbation of COPD and tracheostomy. All-cause mortality will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Omar M Lattouf, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Midtown, Atlanta, Georgia, United States